CLINICAL TRIAL: NCT04569136
Title: Physical Therapy Intervention for Puerperal Mastitis in Breastfeeding Women
Brief Title: Physical Therapy Intervention for Puerperal Mastitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuan-Yin Lin, Assistant professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOST 109-2314-B-006-041-MY3
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-02

CONDITIONS: Mastitis
MeSH Terms: conditions — Mastitis | interventions — Educational Status; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): * Educating the patient about mastitis and self-management strategies
  * Treating with therapeutic ultrasound
  * Administering and teaching breast massage
  Interventions: Other: Education; Other: Therapeutic ultrasound; Other: Breast massage
- Sham group (Sham Comparator): * Educating the patient about mastitis and self-management strategies
  * Receiving sham ultrasound
  * Administering and teaching breast massage
  Interventions: Other: Education; Other: Sham ultrasound; Other: Breast massage
- Usual care group (Other): Receiving usual obstetric care, which may include verbal advice/printed patient information regarding mastitis and breastfeeding from the medical or nursing staff
  Interventions: Other: Usual obstetric care

INTERVENTIONS:
Other: Education — The education session including education about mastitis, feeding techniques, lifestyle changes, thermal/cryo therapy and demonstration of breast self-massage will take approximately 20 minutes.
  Arms: Intervention group; Sham group
Other: Therapeutic ultrasound — Participants will be treated with 5 minutes of therapeutic ultrasound (pulsed mode) at a frequency of 1 Mega Hertz, a duty cycle of 20%, a pulse intensity of 1.8 Watt/centimetre squared. The ultrasound probe will be moved at a speed of about 4 centimetre/second. The intensity and duration will be adjusted if the patient complains of discomfort. The ultrasound transducer head will massage over the tender point on the breast.
  Arms: Intervention group
Other: Sham ultrasound — Participants will receive 5 minutes of 'sham' ultrasound at 0 Watt/centimetre squared intensity from a physical therapist.
  Arms: Sham group
Other: Breast massage — Breast massage includes general and focused massage. Participants will lie in supine position. The breast massage will be applied according to the Vodder method to the affected breast.
  Arms: Intervention group; Sham group
Other: Usual obstetric care — Usual obstetric care may include verbal advice/printed patient information regarding mastitis and breastfeeding from the medical or nursing staff.
  Arms: Usual care group

SUMMARY:
Puerperal mastitis is one of the most commonly reported problems during breastfeeding. Women frequently report breast pain, tenderness, redness, engorgement, fever, malaise, chills, lethargy, sweating, headache, nipple damage and a hot spot on the affected breast. These highly distressing symptoms may severely impact on a woman's daily activities and quality of life and might lead to the premature cessation of exclusive breastfeeding, which may have significant impact on infant health and survival. The role of physical therapy in reducing pregnancy/postpartum-related disorders including breast problems is gaining momentum and importance in obstetrics. However, to date, only low-level evidence has shown positive effects of breast massage, a physical technique, on pain, milk supply and symptom relief in women with breastfeeding problems. This is encouraging, however further research is needed to explore whether physical therapy is effective to reduce symptoms of puerperal mastitis. The investigators will conduct a prospective, assessor blinded single-center randomized controlled trial to assess the effectiveness of an individualized physical therapy program with therapeutic ultrasound, education and massage for patients with puerperal mastitis, compared to patients receiving usual obstetric care and sham ultrasound treatment.

DETAILED DESCRIPTION:
The high incidence of mastitis in breastfeeding women places health professionals working with postpartum women in key positions for managing women for symptoms of mastitis. This study aims to investigate the effectiveness of a physical therapy program for mastitis. The data the investigators collect from this study will provide evidence on effective and targeted strategies to achieve the goals of acceptable, effective and low risk physical therapy treatment of mastitis in postpartum women. Once these perspectives are known, recommendations on mastitis management can be made.

ELIGIBILITY:
Inclusion Criteria:

* Have given birth at National Cheng Kung University Hospital (NCKUH)
* Are Breastfeeding
* Are aged 21-35
* Are diagnosed with early stage mastitis
* Have sufficient Chinese/Mandarin language skills to participate

Exclusion Criteria:

* History of breast reduction or augmentation
* An abscess
* Severe physical/psychiatric impairments
* Presence of any malignancies

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Yin Lin, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diepeveen LC, Fraser E, Croft AJE, Jacques A, McArdle AM, Briffa K, McKenna L. Regional and Facility Differences in Interventions for Mastitis by Australian Physiotherapists. J Hum Lact. 2019 Nov;35(4):695-705. doi: 10.1177/0890334418812041. Epub 2018 Nov 27. PMID 30481473
- [Background] Kasseroller RG. The Vodder School: the Vodder method. Cancer. 1998 Dec 15;83(12 Suppl American):2840-2. doi: 10.1002/(sici)1097-0142(19981215)83:12b+3.0.co;2-5. PMID 9874409
- [Background] Lavigne V, Gleberzon BJ. Ultrasound as a treatment of mammary blocked duct among 25 postpartum lactating women: a retrospective case series. J Chiropr Med. 2012 Sep;11(3):170-8. doi: 10.1016/j.jcm.2012.05.011. PMID 23449233
- [Background] McLachlan Z, Milne EJ, Lumley J, Walker BL. Ultrasound treatment for breast engorgement: A randomised double blind trial. Aust J Physiother. 1991;37(1):23-8. doi: 10.1016/S0004-9514(14)60531-6. PMID 25026196
- [Background] Witt AM, Bolman M, Kredit S, Vanic A. Therapeutic Breast Massage in Lactation for the Management of Engorgement, Plugged Ducts, and Mastitis. J Hum Lact. 2016 Feb;32(1):123-31. doi: 10.1177/0890334415619439. Epub 2015 Dec 7. PMID 26644422
- [Background] Wong RA, Schumann B, Townsend R, Phelps CA. A survey of therapeutic ultrasound use by physical therapists who are orthopaedic certified specialists. Phys Ther. 2007 Aug;87(8):986-94. doi: 10.2522/ptj.20050392. Epub 2007 Jun 6. Erratum In: Phys Ther. 2007 Sep;87(9):1258. PMID 17553923
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Hill PD, Humenick SS. The occurrence of breast engorgement. J Hum Lact. 1994 Jun;10(2):79-86. doi: 10.1177/089033449401000212. PMID 7619260
- [Background] Lim AR, Song JA, Hur MH, Lee MK, Lee MS. Cabbage compression early breast care on breast engorgement in primiparous women after cesarean birth: a controlled clinical trial. Int J Clin Exp Med. 2015 Nov 15;8(11):21335-42. eCollection 2015. PMID 26885074
- [Background] Geissler NJ. An instrument used to measure breast engorgement. Nurs Res. 1967 Spring;16(2):130-6. No abstract available. PMID 5181912
- [Background] Mori H, Uemura N, Koga H, Okazaki M. Objective assessment of reconstructed breast hardness using a durometer. Breast Cancer. 2018 Jan;25(1):81-85. doi: 10.1007/s12282-017-0791-y. Epub 2017 Jun 23. PMID 28646371
- [Background] Teran CG, Torrez-Llanos J, Teran-Miranda TE, Balderrama C, Shah NS, Villarroel P. Clinical accuracy of a non-contact infrared skin thermometer in paediatric practice. Child Care Health Dev. 2012 Jul;38(4):471-6. doi: 10.1111/j.1365-2214.2011.01264.x. Epub 2011 Jun 8. PMID 21651612
- [Background] Jones E, Dimmock PW, Spencer SA. A randomised controlled trial to compare methods of milk expression after preterm delivery. Arch Dis Child Fetal Neonatal Ed. 2001 Sep;85(2):F91-5. doi: 10.1136/fn.85.2.f91. PMID 11517200
- [Derived] Lin KY, Shao W, Tsai YJ, Yang JF, Wu MH. Physical therapy intervention for breast symptoms in lactating women: a randomized controlled trial. BMC Pregnancy Childbirth. 2023 Nov 14;23(1):792. doi: 10.1186/s12884-023-06114-2. PMID 37964187
- Available data/document: Clinical Study Report: DOI：10.6315/2009.37(4)06 — http://www.airitilibrary.com/Publication/alDetailedMesh?DocID=10253009-200912-201002050027-201002050027-261-268

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: * Educating the patient about mastitis and self-management strategies
  * Treating with therapeutic ultrasound
  * Administering and teaching breast massage
  Education: The education session including education about mastitis, feeding techniques, lifestyle changes, thermal/cryo therapy and demonstration of breast self-massage will take approximately 20 minutes.
  Therapeutic ultrasound: Participants will be treated with 5 minutes of therapeutic ultrasound (pulsed mode) at a frequency of 1 Mega Hertz, a duty cycle of 20%, a pulse intensity of 1.8 Watt/centimetre squared. The ultrasound probe will be moved at a speed of about 4 centimetre/second. The intensity and duration will be adjusted if the patient complains of discomfort. The ultrasound transducer head will massage over the tender point on the breast.
  Breast massage: Breast massage includes general and focused massage. Participants will lie in supine position. The breast massage will be applied according to the Vodder method to the affected breast.
- Sham Group: * Educating the patient about mastitis and self-management strategies
  * Receiving sham ultrasound
  * Administering and teaching breast massage
  Education: The education session including education about mastitis, feeding techniques, lifestyle changes, thermal/cryo therapy and demonstration of breast self-massage will take approximately 20 minutes.
  Sham ultrasound: Participants will receive 5 minutes of 'sham' ultrasound at 0 Watt/centimetre squared intensity from a physical therapist.
  Breast massage: Breast massage includes general and focused massage. Participants will lie in supine position. The breast massage will be applied according to the Vodder method to the affected breast.
Period: Overall Study
Arm/Group | Intervention Group | Sham Group | Usual Care Group
Started | 12 | 12 | 13
Completed | 10 | 12 | 12
Not Completed | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Sham Group | Usual Care Group | Total
Number analyzed (Participants) | 12 | 12 | 13 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (3.3) | 33.6 (3.7) | 34.2 (4.4) | 34.1 (3.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12 | 12 | 13 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (3.4) | 24.1 (3.7) | 24.0 (3.7) | 24.2 (3.5)
Waist-hip ratio [Mean (Standard Deviation); unit: Ratio] | 0.83 (0.04) | 0.82 (0.06) | 0.82 (0.04) | 0.83 (0.04)

OUTCOME MEASURES:

1. Primary Outcome: Breast and Nipple Pain
Description: Breast and nipple pain in the past 24 hours will be assessed using the numerical rating scale (NRS). Participants will be asked to rate her breast pain and nipple pain from 0 to 10 (11 point scale), with 0 indicating no pain and 10 indicating the worst possible pain.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group | Sham Group | Usual Care Group
Number analyzed (Participants) | 12 | 12 | 13
score on a scale | 0 [0 to 0.75] | 0 [0 to 0] | 1 [0 to 2]

2. Secondary Outcome: Severity of Breast Engorgement
Description: The degree of breast engorgement of the left and right breasts will be assessed using a six-point engorgement scale developed by Hill and Humenick. The higher scores indicate more severe breast engorgement (1=soft, no change, 2=slight change, 3=firm, non-tender, 4=firm, beginning tenderness, 5=firm, tender, 6=very firm and very tender).
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group | Sham Group | Usual Care Group
Number analyzed (Participants) | 12 | 12 | 13
score on a scale | 1 [1 to 2] | 1.5 [1 to 2] | 2 [1 to 3]

3. Secondary Outcome: Breast Hardness
Description: The assessor will use a portable durometer to measure the hardness of left and right breasts. The participant will lie in a supine position and the durometer will be placed at 3 cm from both nipples in the 10 o'clock and 2 o'clock positions. The spring-loaded presser is pressed downwards until trigger switch on. Each position will be measured three times and the mean value will be obtained. The values range from 0-100. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention Group | Sham Group | Usual Care Group
Number analyzed (Participants) | 12 | 12 | 13
units on a scale | 5.2 [2.8 to 7.4] | 1.0 [0.2 to 5.9] | 2.3 [1.1 to 3.7]

4. Secondary Outcome: Body and Breast Temperature
Description: Core body and breast temperatures will be measured using a non-contact infrared thermometer on the central part of the forehead and in the area 3 cm from both nipples in the 10 o'clock and 2 o'clock positions, respectively. The temperature of each position will be measured three times and the mean value will be recorded.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: Degrees Celsius
Arm/Group | Intervention Group | Sham Group | Usual Care Group
Number analyzed (Participants) | 12 | 12 | 13
Degrees Celsius | 36.9 [36.7 to 37.3] | 36.7 [36.6 to 37.1] | 37.0 [36.7 to 37.4]

5. Secondary Outcome: Volume of Mother's Milk
Description: The volume of mother's milk will be measured by an electric breast pump for 15 minutes. Milk volumes will be recorded by weighing the collecting bottle on an electronic digital scale to the nearest 0.1 gram before and after each expression.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | Intervention Group | Sham Group | Usual Care Group
Number analyzed (Participants) | 12 | 12 | 13
g | 52.2 [20.6 to 81.5] | 17.8 [2.6 to 35.3] | 40.7 [16.9 to 112.0]

6. Secondary Outcome: Acceptability of the Intervention Program
Description: Acceptability of the intervention program will be assessed immediately post-intervention using a short questionnaire with 5-point Likert scale response to questions of 'how acceptable did you find the physical therapy interventions used in this study?' and 'how would you rate your overall satisfaction with the physical therapy program?' from 1 to 5, with 1 indicating very low acceptability or satisfaction and 5 indicating very high acceptability or satisfaction. The number of participants who rate a 5 (i.e. very high) on acceptability and satisfaction will be counted and recorded.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Sham Group | Usual Care Group
Number analyzed (Participants) | 12 | 12 | 13
Participants | 11 | 11 | 7

7. Secondary Outcome: Number of Participants Reporting Adverse Events
Description: Adverse events will be recorded and reported as per Institutional Review Board, National Cheng Kung University Hospital guidelines on reporting adverse events and serious adverse events, with the absence of adverse or serious adverse events related to the physical therapy intervention used to indicate safety of the trial protocol.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Sham Group | Usual Care Group
Number analyzed (Participants) | 12 | 12 | 13
Participants | 0 | 0 | 0

8. Secondary Outcome: Breastfeeding Self-efficacy
Description: Breastfeeding self-efficacy will be evaluated using the Breastfeeding Self-Efficacy Scale - Short Form (BSES-SF). The BSES-SF is a validated and reliable patient-reported outcome measure consisting of 14 items. Each item is scored between 1-5 points with 1 indicating 'not at all confident' and 5 indicating 'always confident'. Total scores range from 14 to 70, with higher scores indicating higher breastfeeding self-efficacy.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group | Sham Group | Usual Care Group
Number analyzed (Participants) | 12 | 12 | 13
score on a scale | 52.0 [40.0 to 58.0] | 59.5 [34.25 to 68.75] | 55 [52.5 to 59.5]

ADVERSE EVENTS:
Time Frame: 2 years
Description: The definition of adverse event and serious adverse event, used to collect adverse event information, is the same as those from the clinicaltrials.gov Definitions.
Arm/Group | Intervention Group | Sham Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT04569136/Prot_SAP_000.pdf